CLINICAL TRIAL: NCT01417910
Title: Prognostic Markers of Outcome in Patients Undergoing Infra-inguinal Revascularisation. A Prospective Observational Study.
Brief Title: Predictors of Post Operative Outcome in Peripheral Vascular Surgical Patients
Status: Completed | Type: Observational
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PVD10
Record Dates: First submitted 2011-08-01; First posted 2011-08-16 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-02

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral vascular disease: Subjects who have peripheral vascular disease

SUMMARY:
Over 3000 people each year undergo bypass operations to their lower limbs, and these operations carry significant risks with approximately 1 in 20 of these people dying in hospital, and another 1 in 20 having a heart attack.

Assessment of these patients in order to stratify their risk of both dying and having significant complications aid in improving their care, enable better utilisation of scarce critical care resources, and allow us to give patients better information on which to base consent.

Aims The aims of the project are to assess the feasibility of exercise testing this group of patients both with cycle and arm exercise, and to identify markers of outcome in this group.

Methodology This is a prospective observational study designed to test the hypothesis that a combination of cardiopulmonary exercise testing and blood tests provides prognostic value on outcome measures after surgery for lower limb revascularisation

Subjects will have 2 exercise tests, one arm and one cycle, prior to surgery at their preoperative assessment appointment. From these tests we will measure how much work patients can do, how much oxygen they are able to use, and when the heart is unable to deliver enough oxygen to the cells. In addition they will have blood samples taken prior to the operation (brain natriuretic peptide), and on days 1 and 3 (troponin I) after the operation to look at cardiac markers of damage.

This data will be used to see if we can predict those patients that have both short and long term complications, and also to see whether the different forms of exercise testing are comparable, or if one type is superior.

Expected outcomes We expect that through a combination of exercise testing and blood test we will be able to identify patients at increased risk of complications after surgery. We also expect to find that arm exercise will be a more feasible and informative test that cycle exercise.

DETAILED DESCRIPTION:
Background Over 3000 people each year undergo bypass operations to their lower limbs, and these operations carry significant risks with approximately 1 in 20 of these people dying in hospital, and another 1 in 20 having a heart attack. The number of people having this type of procedure has grown over recent years and the trend is predicted to continue. Due to this significant increase in the volume of these patients, and the associated complications that occur with this surgery, utilisation of more resources such as critical care is often needed.

Assessment of these patients in order to stratify their risk of both dying and having significant complications aid in improving their care, allow better utilisation of scarce critical care resources, and also allow us to provide patients with better information as part of the informed consent process.

A high risk group in major abdominal surgery can be identified through a simple exercise test (cardiopulmonary exercise test) that looks at how the body uses oxygen, and also through a blood test that look at a hormone secreted by the heart. Vascular surgical patients are at risk for the development of major cardiac complications in the postoperative period but a system for appropriate preoperative risk stratifications has yet to be achieved.

Aims The aims of the project are to assess the feasibility of exercise testing this group of patients both with cycle and arm exercise, and to identify markers of outcome in this group. Identification of markers that can predict how patients will fare after surgery will allow us to improve the informed consent process, utilise resources more effectively and efficiently and identify opportunities to attempt to modify outcomes.

Methodology This is a prospective observational study designed to test the hypothesis that a combination of cardiopulmonary exercise testing and blood tests provide prognostic value on outcome measures after surgery for lower limb revascularisation.

Participants will have 2 exercise tests, one arm and one cycle, prior to surgery at their preoperative assessment appointment. From these tests we will measure how much work patients can do, how much oxygen they are able to use, and when the heart is unable to deliver enough oxygen to the cells. In addition they will have blood samples taken prior to the operation (brain natriuretic peptide), and on days 1 and 3 (troponin I) after the operation to look at cardiac markers of damage.

This data will be used to see if we can predict those patients that have both short and long term complications, and also to see whether the different forms of exercise testing are comparable, or if one type is superior.

Expected outcomes We expect that through a combination of exercise testing and a blood test we will be able to identify patients at increased risk of complications after surgery. We also expect to find that arm exercise will be a more feasible and informative test that cycle exercise.

Implications Identification of a high risk group would allow appropriate strategies to be implemented to reduce risk, and allow better post-operative resource utilisation. This study will also allow a larger multicentre study to be adequately powered and constructed.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective and expedited infra inguinal peripheral revascularisation. Patients undergoing radiological assessment (angiography) and/or radiological intervention for peripheral vascular disease

Exclusion Criteria:

* Patients refusing to participate in the study or unable to give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with peripheral vascular disease in a secondary care setting scheduled to undergo infra inguinal revascularisation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
1 year all cause mortality | 1 year

SECONDARY OUTCOMES:
1 year major adverse cardiac event. | 1 year
Morbidity as measured by the Post operative morbidity survey | 7 days
major adverse cardiac event. | participants will be followed for the duration of hospital stay, an expected median of 10 days
30 day all cause mortality. | 30 day
Surgical post operative complications | participants will be followed for the duration of hospital stay, an expected median of 10 days
  participants will be followed for the duration of hospital stay, an expected median of 10 days
Medical post operative complications | participants will be followed for the duration of hospital stay, an expected median of 10 days
  participants will be followed for the duration of hospital stay, an expected median of 10 days
Quality of life measured at 6 and 12 months postoperatively by the EQ-5D-5L questionnaire. | 0,6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Davies, MBChB, Principal Investigator — York Teaching Hospital NHS Foundation Trust
Locations (1):
- York Teaching Hospitals NHS Foundation Trust, York, North Yorkshire, United Kingdom